CLINICAL TRIAL: NCT01665391
Title: A Phase 2, Multicenter, Double-Blind, Parallel Dosing, Randomized Study of Fresolimumab or Placebo in Patients With Steroid-Resistant Primary Focal Segmental Glomerulosclerosis
Brief Title: A Study of Fresolimumab in Patients With Steroid-Resistant Primary Focal Segmental Glomerulosclerosis (FSGS)
Acronym: FSGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC1008FSGS03110; 2010-019545-25 (EudraCT Number); U1111-1139-9082 (Other: World Health Organization Universal Trial Number (UTN)); DRI12792 (Other: Sanofi)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Primary Focal Segmental Glomerulosclerosis
MeSH Terms: interventions — fresolimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fresolimumab 1 mg/kg total body weight (Experimental)
  Interventions: Drug: fresolimumab
- fresolimumab 4 mg/kg total body weight (Experimental)
  Interventions: Drug: fresolimumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fresolimumab — 1 mg/kg total body weight administered intravenous (IV)
  Arms: fresolimumab 1 mg/kg total body weight
Drug: fresolimumab — 4 mg/kg total body weight administered intravenous (IV)
  Arms: fresolimumab 4 mg/kg total body weight
Drug: Placebo — Placebo administered to match active treatment group
  Arms: Placebo

SUMMARY:
The primary objectives of this trial are as follows:

* to compare the achievement of a partial remission (PR) or complete remission (CR) in urinary protein: creatinine ratio (Up/c ratio) in patients treated with fresolimumab versus placebo
* to compare the safety profile of patients treated with fresolimumab versus placebo

The secondary objectives are as follows:

* To compare the reduction in proteinuria in patients treated with fresolimumab versus placebo
* To evaluate fresolimumab dose-dependent reduction in proteinuria
* To compare the change in renal function (estimated glomerular filtration rate [eGFR]) in patients treated with fresolimumab versus placebo
* To evaluate the multiple-dose pharmacokinetics of fresolimumab

ELIGIBILITY:
Inclusion Criteria:

* The patient's renal biopsy is consistent with the diagnosis of primary Focal Segmental Glomerulosclerosis (FSGS) including all histological subtypes.
* The patient has an eGFR ≥ 30 mL/min/1.73 m2
* The patient has a urinary total protein:creatinine ratio ≥ 3 mg protein/mg creatinine
* In the opinion of the Investigator, the patient has steroid-resistant FSGS. The patient must have been treated for FSGS with a course of high-dose steroid therapy for a minimum of 4 weeks
* The patient has been treated with an ACEi (angiotensin converting enzyme inhibitor) and/or ARB (angiotensin receptor blocker) at a stable dose for a minimum of 4 weeks prior to Visit 2 (treatment start)

Exclusion Criteria:

* The patient has FSGS which in the Investigator's opinion is secondary to another condition
* The patient has been taking prednisone at a dose > 10 mg/day (or equivalent dose of an alternative glucocorticoid) within 4 weeks prior to Visit 1 (Screening Visit).
* The patient has received any other systemically administered immunosuppressive drugs (other than glucocorticoids) within 8 weeks prior to Visit 1.
* The patient has received rituximab within 6 months prior to Visit 1.
* The patient has a history of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving partial remission (PR) or complete remission (CR) in urinary protein: creatinine ratio (Up/c ratio) | Up to Day 112
Number of patients reporting adverse events (AEs), serious adverse events (SAEs), and medical events of interest (MEOIs) | Up to Day 112

SECONDARY OUTCOMES:
Percentage of patients achieving CR in Up/c ratio | Up to Day 112
Percentage of patients achieving PR in Up/c ratio | Up to Day 112
Change from baseline in Up/c ratio and urinary protein excretion rate | Up to Day 112
Time to first PR or CR | Up to Day 112
Change from baseline in eGFR (estimated glomerular filtration rate) | Up to Day 112
Percentage of patients achieving PR or CR with stable eGFR (estimated glomerular filtration rate) | Up to Day 112
Mean Fresolimumab serum concentration at each sample collection time point | Up to Day 252

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (32):
- United States (21):
  - Investigational Site Number 4008, Birmingham, Alabama
  - Investigational Site Number 4029, Phoenix, Arizona
  - Investigational Site Number 4009, San Francisco, California
  - Investigational Site Number 4023, Stanford, California
  - Investigational Site Number 4005, Atlanta, Georgia
  - Investigational Site Number 4019, Springfield, Illinois
  - Investigational Site Number 4004, Baltimore, Maryland
  - Investigational Site Number 4002, Bethesda, Maryland
  - Investigational Site Number 4022, Boston, Massachusetts
  - Investigational Site Number 4012, Ann Arbor, Michigan
  - Investigational Site Number 4025, Detroit, Michigan
  - Investigational Site Number 4006, Rochester, Minnesota
  - Investigational Site Number 4024, St Louis, Missouri
  - Investigational Site Number 4016, New York, New York
  - Investigational Site Number 4003, New York, New York
  - Investigational Site Number 4014, Rosedale, New York
  - Investigational Site Number 4018, Philadelphia, Pennsylvania
  - Investigational Site Number 4001, Chattanooga, Tennessee
  - Investigational Site Number 4020, Dallas, Texas
  - Investigational Site Number 4027, Houston, Texas
  - Investigational Site Number 4013, Seattle, Washington
- Investigational Site Number 4104, Porto Alegre, Brazil
- Germany (3):
  - Investigational Site Number 4302, Aachen
  - Investigational Site Number 4301, Düsseldorf
  - Investigational Site Number 4304, Hamburg
- Italy (4):
  - Investigational Site Number 4401, Bari
  - Investigational Site Number 4404, Bergamo
  - Investigational Site Number 4403, Montichiari
  - Investigational Site Number 4405, Reggio Calabria
- Spain (3):
  - Investigational Site Number 4503, Barcelona
  - Investigational Site Number 4504, Madrid
  - Investigational Site Number 4502, Madrid

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732